CLINICAL TRIAL: NCT05902416
Title: Clinical Registration Study of Haploidentical Stem Cell Transplantation for Elderly Patients With Acute Leukemia or Myelodysplastic Syndrome
Brief Title: Clinical Registration Study of Haplo-HSCT for Elderly Patients With Acute Leukemia/ Myelodysplastic Syndrome
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Principal Investigator, Peking University People's Hospital
Other Study IDs: 2022PHB352-001
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Leukemia; Myelodysplastic Syndromes
Keywords: RIC regimen; Elderly; comorbidity; transplant-related mortality; Haplo-HSCT
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RIC regimen,Elderly,Haplo-HSCT,PFS,OS,TRM

SUMMARY:
This study is an open, prospective, single-center, single-arm study expanded based on the study of NCT03412409.The primary objective of this study is to evaluate the transplantation efficacy of the RIC conditioning regimen in elderly patients receiving the transplantation of haploidentical hematopoietic stem cells. Elderly patients are defined as ≥55 years of age; High comorbidity is defined as an HCT-CI score ≥3.Primary endpoint is 1-year LFS. Secondary endpoints are 1-year OS and 1-year TRM, Other indicators to be assessed in this study include acute GVHD, chronic GVHD, CMV activation, EBV activation, engraftment.

DETAILED DESCRIPTION:
Currently, the transplantation of allogeneic hematopoietic stem cells (allo-SCT) remains the main and often the only cure for neoplastic hematologic disorder or hematological malignancy. Although HLA-matched siblings are the preferred donor, not all patients have one; or it needs to wait so long to obtain it that the optimal time for transplantation is past. Haploidentical transplants as secondary donors are more readily available and may be considered in combination with the conditions of the donor and the patient and the experience of the transplant facility when a matched donor is unavailable. Currently, haploidentical transplantation has been commonly applied to young patients. On the other hand, TRM rate will be higher in elderly patients and patients with high comorbidity due to tolerability, thus reducing the ultimate benefits of patients.

The choice of conditioning regimen is influenced by multiple factors such as disease type, disease status, physical condition, and source of transplant donor. For patients over 55 years of age or with a comorbidity index ≥3, the RIC regimen may be considered to improve patient tolerability. RIC regimen can improve the tolerability of patients receive transplants, while regimens such as immune suppressants are also needed to control and improve the overall transplant efficiency. An in-depth study of RIC regimen will help improve the effects of transplantation and increase patient benefits.

This study is aim to evaluate the efficacy of RIC conditioning regimen for transplantation in elderly patients or patients with high comorbidity receiving the transplantation of haploidentical hematopoietic stem cells.

Drugs and dosage of conditioning regimen:

Ara-C(2g/m2/day,-10 days to -9 days),Bu(9.6mg/kg,-8 days to -6 days),Flu(30mg/m2/day,-6 days to -2 days),Cy(1,000mg/m2/day,-5 days to -4 days),semustine(250mg/m2,-3 days),ATG(10 mg/kg,-5 to -2 days).

Supportive care:

CsA: To prevent GVHD, CsA therapy starts 9 days before transplantation at 2.5 mg/kg intravenously until gut function returns to normal after transplantation; CsA is then orally administered. MMF: To prevent GVHD, 0.5g of MMF is orally administered every 12 hours 9 days before transplantation until hematopoietic function is restored after transplantation. MTX: To prevent GVHD, MTX is intravenously administered at 15 mg/m2 on day 1 after transplantation. On days 3, 6 and 11 after transplantation, MTX is intravenously administered at 10 mg/m2. Ganciclovir: To prevent post-transplantation CMV infection, it is administered 2 days before transplantation, and to prevent post-transplantation CMV infection, it is orally administered at 400 mg twice a day until the end of all immunosuppressive medications.

Primary endpoint is 1-year LFS. Secondary endpoints are 1-year OS and 1-year TRM, Other indicators to be assessed in this study include acute GVHD, chronic GVHD, CMV activation, EBV activation, engraftment.

CMV and EBV Tests are performed twice weekly for monitor based on PCR means.

The follow-up period designed for this study is 1 year, with the day of hematopoietic stem cell transplantation as Day 1 and the visit dates of Day 0, 1st month, 2nd month, 3rd month, 6th month and 12th month. The end of the study is defined as the date of the last visit of the last patient (LPLV).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥55 years of age and <70 years of age, with acute leukemia or MDS (with or without HCT-CI≥3);
* Patients eligible for the transplantation of allogeneic hematopoietic stem cells;
* Patients unavailable with HLA matched donors but available with haploidentical donors;
* Voluntary participation in this study and signing the informed consent form.

Exclusion Criteria:

* Patients with the severe infections;
* Pregnant or lactating women or female and male subjects of childbearing age and their spouses who are unable to secure effective contraception during the dosing period and within 90 days after the end of the dosing period.
* Patients who are not eligible for hematopoietic stem cell transplantation;
* Patients who are enrolled in other clinical trials within 1 month;
* Patients who may not be able to complete the study for other reasons, or may be considered by the investigator not suitable to participate in the study;
* Patients unable to properly understand or refusing to accept the informed consent form.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥55 years of age and <70 years of age, with acute leukemia or MDS (with or without HCT-CI≥3)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
1-year LFS | Participants will be followed for an expected average of 1 years
  defined as disease relapse, disease progression or death (whichever occurs first) within 1 year from the day the patient receives transplantation.

SECONDARY OUTCOMES:
1-year OS | Participants will be followed for an expected average of 1 years
  defined as survival rate within 1 year from the day the patient receives transplantation, calculated based on death from any cause.
1-year TRM | Participants will be followed for an expected average of 1 years
  defined as death from any cause other than disease relapse within 1 year from the day the patient receives transplantation.

OTHER OUTCOMES:
Adverse event | Participants will be followed for an expected average of 1 years
  The incidence rate of acute GVHD, chronic GVHD, CMV activation, EBV activation after transplantation
Engraftment rate | Participants will be followed for an expected average of 1 years
  The success rate of engraftment after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes